CLINICAL TRIAL: NCT00885677
Title: MOnitoring REsynchronization deviCes and cARdiac patiEnts
Acronym: MORE-CARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDT-MORE-CARE
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): Patients of the study arm are CRT-D patients followed-up by means of a remote disease management system (Medtronic Carelink® Network), for which an automatic alerting system is enabled for fluid accumulation, AT/AF episodes and system integrity.
  Interventions: Device: Medtronic CareLink® Network
- Control Group (No Intervention): Patients are CRT-D patients managed according to current standard clinical practice, based on routinely performed in-office visits.

INTERVENTIONS:
Device: Medtronic CareLink® Network — Continuous monitoring via a disease remote management system.
  Patients of the Study group will receive a remote monitor and their device will be programmed to have wireless telemetry, Care Alerts, and the ability to transmit over the Medtronic CareLink® network. Clinical and device conditions will be then monitored continuously and alarms for the physician will be generated if a set of pre-defined potentially harming conditions should occur.
  Arms: Study Group

SUMMARY:
The objective of this study is to compare two different strategies of disease management in heart failure patients treated with cardiac resynchronization therapy devices

1. Remote monitoring with CareLink Network System
2. Standard management of the disease by means of scheduled routine in-patient follow-ups;

and to demonstrate that the remote monitoring strategy is superior to the standard strategy, both in terms of clinical effectiveness and total healthcare system utilization.

DETAILED DESCRIPTION:
Major cardiovascular adverse events in patients with heart failure treated with cardiac resynchronization therapy (CRT-D) represent a big concern to the medical community, as they require hospitalizations and may lead to death.

Subjects with a history of heart failure are counseled regarding the importance of contacting their clinicians promptly if they experience any changes or worsening of their condition.

Acute heart failure episodes with hospitalizations represent one of the most relevant causes of health status deterioration for these patients. Moreover, atrial arrhythmias occurrence is a big issue, as it increases the risk of heart failure itself, stroke and inappropriate shocks. In addition to affecting patient health, hospital admission resulting from these complications will impact healthcare costs.

Latest generations of Medtronic CRT-D devices are equipped with a system that triggers an alarm if possible fluid accumulation is detected (OptiVol). This may initiate patient-clinician contact before evident cardiac decompensation. Moreover, advanced diagnostic capabilities for detecting atrial arrhythmias occurrence and total burden are available on such devices.

Importantly, all these devices are now able to inform physician of these events by remote monitoring with CareLink Network parameters, and have the potential of playing a key role in patient monitoring.

Over the last years, interest has been increasing in remote monitoring models for delivering care to HF patients, either as telemonitoring (transfer of physiological data through telephone or digital cable from home to healthcare provider) or as regular structured telephone contacts between patients and healthcare providers, which may or may not include data transfer.

Several studies with relatively large numbers of patients have been published (see table).

A recent meta-analysis found that remote monitoring programs for patients with chronic HF living in the community reduced admissions to hospital and all cause mortality by nearly one fifth while improving health related quality of life, but had no significant effect on all cause admission to hospital.

However, none of the published studies considered remote monitoring systems able to provide device-detected information on fluid accumulation, AT/AF total burden, arrhythmias occurrence and device-related issues in patients treated with CRT-D devices.

Early intervention may then be a key element in avoiding major cardiovascular events to occur and possible deterioration of the disease progression. The Carelink Network remote monitoring system, through Care Alerts, may initiate subject-clinician contact before typical signs and symptoms are exhibited, since it provides the physician with an automatic alert for atrial arrhythmias occurrence, fluid accumulation, and system integrity issues. However, clinical evidence must be provided of the superiority of this patient management strategy with respect to standard clinical practice, based on routine in-office visits.

Very recent findings showed that the use of CareLink in European clinical practice is technically feasible and that remote follow-up is an efficient method of surveillance of implanted patients. Moreover, the early detection and review of device and clinical events suggest the potential impact of remote monitoring on overall patient care.

There are a number of possible limitations with remote monitoring. The CareLink Network system requires that the patient establishes an initial contact between the device and the remote monitor unit, and that the unit is properly hooked up to the phone line. Not all patients may be able to perform the setup properly. There may be a delay by the physician in consulting patient data (for example over weekends), with a risk of adverse events occurring during that interval. There may be difficulties in contacting patients (e.g. if they are traveling). These possible limitations need to be properly assessed, especially for monitoring atrial arrhythmias, where the time factor is of importance for avoiding complications.

Remote patients' disease management has the potential for avoiding hospitalization. Clear demonstration that remote monitoring of AT/AF/HF plus strict treatment guidelines leads to a reduction in hospitalization rates has not been proven, and it could be a major argument for using this technology in routine clinical practice.

The MORE-CARE Study is aimed at comparing two different strategies of disease management in heart failure patients treated with CRT-D devices:

1. Remote disease management via Carelink Network system
2. Standard disease management by means of scheduled routine in-patient follow-ups. The main objective of the study is to demonstrate that the remote management strategy is superior to the standard strategy, both in terms of clinical effectiveness and total healthcare system utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated to CRT-ICD according to current guidelines:
* Left ventricular systolic dysfunction (LVEF≤35%),
* New York Heart Association functional class III-IV,
* QRS≥120 ms
* Optimized medical treatment.
* Patient implanted within the last 8 weeks with Medtronic CRT-ICD device equipped with fluid accumulation diagnostics, AT/AF monitoring capability, wireless telemetry for automatic remote data transmission and alerting system for physician.
* Patient with less than 8 weeks follow-up, who has not received Carelink® Network Monitor and was not managed by Cardiac Compass report reviewing.
* Carelink Network is available at patient's home
* Patient or the patient's caregiver is willing and able to use the Medtronic CareLink® Network Monitor and to perform the required duties at home or has a family member or assistant perform those duties.
* Patient is willing and able to sign an informed consent form.

Exclusion Criteria:

* Inability to fully understand the instructions relating to remote monitoring using CareLink® Network.
* Permanent AT/AF.
* Patient had not been previously implanted with a CRT/CRT-D device.
* Patient has medical conditions that would limit study participation.
* Patient is less than 18 years of age.
* Patient is enrolled in or intends to participate in another clinical trial that may have an impact on the study endpoints.
* Patient meets any exclusion criteria required by local law.
* Inability or refusal to sign a patient informed consent form.
* Patient's life expectancy is less than one year in the opinion of the physician
* Patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2009-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haran Burri, MD, Principal Investigator — University Hospitals of Geneva Switzerland; Giuseppe Boriani, MD, Principal Investigator — Policlinico Universitario Sant'Orsola, Bologna, Italy; Renato Pietro Ricci, MD, Principal Investigator — Azienda Ospedaliera San Filippo Neri, Roma, Italy; Aurelio Quesada, MD, Principal Investigator — Hospital General Universitario de Valencia, Spain; Stefano Favale, MD, Principal Investigator — Policlinico Universitario di Bari, Italy; Josef Kautzner, MD, Principal Investigator — IKEM, Prague, Czech Republic; Antoine Da Costa, MD, Principal Investigator — Hopital du Nord, Saint Etienne, France
Locations (64):
- Institut Klinicke a Experimentalni Mediciny, Prague, Czechia
- France (12):
  - Centre Hospitalier Universitaire de Angers, Angers
  - Hôpital Cardiologique du Haut Lévêque, Bordeaux
  - Centre Hospitalier, La Rochelle
  - Hopital Louis Pradel, Lyon
  - Hopital Saint Joseph, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU, Narbonne
  - Hopital La Source, Orléans
  - Hopital La Pitie Salpetriere, Paris
  - Clinique Bizet, Paris
  - Hopital du Nord, Saint-Etienne
  - CHRU, Tours
- Greece (5):
  - Evaggelismos Hospital, Athens
  - Henry Dynant Hospital - Athens, Athens
  - University Hospital Herakleion, Heraklion
  - HYGEIA - Hospital, Marousi
  - University Hospital AHEPA Thessaloniki, Thessaloniki
- Hungary (2):
  - Gottsegen György Országos Kardiológia Intézet GOKI, Budapest
  - Semmelweis University AOK, Budapest
- Wolfson Medical Center, Holon, Israel
- Italy (29):
  - Ospedale Civile, Chioggia, Venezia
  - Ospedale Civile, Mirano, Venezia
  - Policlinico Universitario, Bari
  - Cliniche Gavazzeni, Bergamo
  - Ospedali Riuniti, Bergamo
  - Policlinico Universitario S. Orsola-Malpighi, Bologna
  - Fondazione Poliambulanza, Brescia
  - Ospedale V.E. Ferrarotto, Catania
  - Ospedale Pugliese e Ciaccio, Catanzaro
  - Sant'Anna Hospital, Catanzaro
  - Ospedale Unico della Versilia, Lido Di Camaiore (LU)
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Paolo, Milan
  - A.O. Monaldi, Napoli
  - Azienda Ospedaliera Sacro Cuore Don Calabria, Negrar
  - Ospedale Giovan Battista Grassi, Ostia Antica
  - Clinica San Carlo, Paderno Dugnano
  - Ospedali Civico e Benfratelli, Palermo
  - Ospedale San Salvatore, Pesaro
  - Istituto di Fisiologia Clinica - CNR, Pisa
  - Ospedale Santa Maria delle Croci, Ravenna
  - Azienda Complesso Ospedaliero San Filippo Neri, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - Ospedale Santa Maria Del Carmine, Rovereto
  - P.O. di Trento P.O.S.Chiara, Trento
  - Azienda Ospedaliera-Ospedali Riuniti, Trieste
  - Ospedale E. Macchi, Varese
  - Ospedale Civile Maggiore di Borgo Trento, Verona
- MC Haaglanden - Locatie Westeinde, The Hague, Netherlands
- Slovakia (2):
  - NUSCH, Bratislava
  - VUSCH, Košice
- Spain (7):
  - Hospital De Torrevieja, Alicante
  - Hospital Reina Sofia, Córdoba
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario de Valme, Seville
  - Hospital General Universitario, Valencia
  - Hospital Universitario La Fé, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Switzerland (4):
  - Universitätsspital, Basel
  - University Hospital, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - Triemli Hospital, Zurich

REFERENCES:
- [Background] Burri H, Quesada A, Ricci RP, Boriani G, Davinelli M, Favale S, Da Costa A, Kautzner J, Moser R, Navarro X, Santini M. The MOnitoring Resynchronization dEvices and CARdiac patiEnts (MORE-CARE) study: rationale and design. Am Heart J. 2010 Jul;160(1):42-8. doi: 10.1016/j.ahj.2010.04.005. PMID 20598971
- [Result] Boriani G, Da Costa A, Ricci RP, Quesada A, Favale S, Iacopino S, Romeo F, Risi A, Mangoni di S Stefano L, Navarro X, Biffi M, Santini M, Burri H; MORE-CARE Investigators. The MOnitoring Resynchronization dEvices and CARdiac patiEnts (MORE-CARE) randomized controlled trial: phase 1 results on dynamics of early intervention with remote monitoring. J Med Internet Res. 2013 Aug 21;15(8):e167. doi: 10.2196/jmir.2608. PMID 23965236
- [Derived] Burri H, da Costa A, Quesada A, Ricci RP, Favale S, Clementy N, Boscolo G, Villalobos FS, Mangoni di S Stefano L, Sharma V, Boriani G; MORE-CARE Investigators. Risk stratification of cardiovascular and heart failure hospitalizations using integrated device diagnostics in patients with a cardiac resynchronization therapy defibrillator. Europace. 2018 May 1;20(5):e69-e77. doi: 10.1093/europace/eux206. PMID 28679168
- [Derived] Boriani G, Da Costa A, Quesada A, Ricci RP, Favale S, Boscolo G, Clementy N, Amori V, Mangoni di S Stefano L, Burri H; MORE-CARE Study Investigators. Effects of remote monitoring on clinical outcomes and use of healthcare resources in heart failure patients with biventricular defibrillators: results of the MORE-CARE multicentre randomized controlled trial. Eur J Heart Fail. 2017 Mar;19(3):416-425. doi: 10.1002/ejhf.626. Epub 2016 Aug 28. PMID 27568392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 918 patients have been enrolled in the study, from 29/05/2009 (date of first enrollment) until 20/08/2014 (date of last enrollment).
Pre-assignment Details: 918 subjects signed the Informed Consent Form. One of those subjects withdraw from the study prior randomization, therefore 917 subjects were randomized either to Study (462) or to Control (455) groups.
Groups:
- Study Group: Patients of the study arm are CRT-D patients followed-up by means of a remote disease management system (Medtronic Carelink® Network), for which an automatic alerting system is enabled for fluid accumulation, AT/AF episodes and system integrity.
  Medtronic CareLink® Network: Continuous monitoring via a disease remote management system.
  Patients of the Study group will receive a remote monitor and their device will be programmed to have wireless telemetry, Care Alerts, and the ability to transmit over the Medtronic CareLink® network. Clinical and device conditions will be then monitored continuously and alarms for the physician will be generated if a set of pre-defined potentially harming conditions should occur.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 462 | 455
Intention To Treat | 437 | 428
Completed | 279 | 277
Not Completed | 183 | 178
Not completed — Death | 40 | 34
Not completed — Lost to Follow-up | 15 | 13
Not completed — Protocol Violation | 54 | 54
Not completed — premature study closure | 41 | 44
Not completed — device/lead revision or replacement | 7 | 6
Not completed — Heart transplantation | 1 | 0
Not completed — Inclusion/exclusion not met | 25 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 437 | 428 | 865
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 67 (10) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 116 | 211
  Male | 342 | 312 | 654
Region of Enrollment [Number; unit: participants]
  Greece | 21 | 19 | 40
  Netherlands | 4 | 5 | 9
  Hungary | 6 | 6 | 12
  Italy | 225 | 231 | 456
  Israel | 3 | 3 | 6
  Slovakia | 12 | 11 | 23
  France | 85 | 77 | 162
  Switzerland | 35 | 33 | 68
  Spain | 46 | 43 | 89
History of AF [Number; unit: participants]
  History of AF | 89 | 62 | 151
  No History of AF | 340 | 361 | 701
  Missing | 8 | 5 | 13
History of Myocardial Infarction [Number; unit: participants]
  With History of Myocardial Infarction | 164 | 173 | 337
  Without History of Myocardial Infarction | 262 | 252 | 514
  Missing | 11 | 3 | 14
LVEF [Mean (Standard Deviation); unit: %] | 27.3 (6.6) | 27.4 (6.0) | 27.3 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Median Time Between Event Onset Time and Clinical Decision for Each Subject.
Description: The median delay from device-detected events to clinical decisions was considerably shorter in the Remote group compared to the Control group
Time Frame: 1 year since the randomization
Population: Phase 1: A total of 154 patients were enrolled from May 2009 through April 2010 from 32 centers in 6 different countries (France, Hungary, Israel, Italy, Spain, and Switzerland). The final patient cohort object of analysis comprised 148 patients (76 in the Remote group and 72 in the Control group)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 76 | 72
days | 2 [1 to 4] | 29 [3 to 51]

2. Primary Outcome: Phase 2: Combined Endpoint of Death From Any Cause, Cardiovascular and Device-related Hospitalizations (at Least 48 Hours Stay), Calculated as Number of Subjects With at Least One Event
Description: Time to first event
Time Frame: 2 years after randomization
Population: All subjects in analysis were included in the primary endpoint analysis
Measure: Number; unit: participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 437 | 428
participants | 134 | 126

ADVERSE EVENTS:
Time Frame: Adverse events have been collected since subject enrollment until subjct exit/death.
Description: The following Serious Adverse Events and Adverse Device Effects needed to be reported to Medtronic:
  * Serious Adverse Events (SAE);
  * Serious Adverse Device Effects (SADE);
  * Serious Adverse Procedure related Events (SAPE);
  * Unexpected Serious Adverse Effects (USAE). (Definition ISO EN ISO 14155-1)
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 184/462 | 168/455
Other Adverse Events (participants affected / at risk) | 68/462 | 85/455
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=462) | Control Group (N=455)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 3 (6) | 2 (2)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Cardiac disorders) | 10 (12) | 11 (11)
Cardiac arrhythmias (Cardiac disorders) | 16 (22) | 19 (21)
Cardiac disorder signs and symptoms (Cardiac disorders) | 16 (16) | 12 (14)
Cardiac valve disorders (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery disorders (Cardiac disorders) | 1 (1) | 4 (4)
Heart failures (Cardiac disorders) | 76 (132) | 73 (133)
Myocardial disorders (Cardiac disorders) | 0 (0) | 1 (1)
Surgical and medical procedures (Cardiac disorders) | 1 (1) | 2 (2)
Vascular disorders (Cardiac disorders) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (2) | 3 (3)
Anterior eye structural change, deposit and degeneration (Eye disorders) | 2 (3) | 1 (1)
Abdominal hernias and other abdominal wall conditions (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal haemorrhages NEC (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatal outcome (General disorders) | 21 (21) | 20 (20)
General system disorders NEC (General disorders) | 7 (7) | 8 (9)
Tissue disorder (General disorders) | 1 (1) | 0 (0)
Tissue disorders NEC (General disorders) | 0 (0) | 1 (2)
Gallbladder disorders (Hepatobiliary disorders) | 2 (2) | 0 (0)
Infections - pathogen unspecified (Infections and infestations) | 2 (2) | 2 (2)
Infections and infestations (Infections and infestations) | 4 (4) | 4 (4)
Bone and joint injuries (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Cardiac disorder signs and symptoms (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Medication errors (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural and device related injuries and complications NEC (Injury, poisoning and procedural complications) | 32 (33) | 26 (28)
Cardiac and vascular investigations (excl enzyme tests) (Investigations) | 2 (2) | 1 (1)
Gastrointestinal investigations (Investigations) | 1 (1) | 0 (0)
Diabetic complications (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (2)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 8 (9)
Central nervous system vascular disorders (Nervous system disorders) | 3 (3) | 4 (4)
Headaches (Nervous system disorders) | 1 (1) | 0 (0)
Increased intracranial pressure and hydrocephalus (Nervous system disorders) | 1 (1) | 1 (2)
Neurological disorders NEC (Nervous system disorders) | 5 (5) | 0 (0)
Renal disorders (excl nephropathies) (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disturbances (incl subtypes) (Nervous system disorders) | 0 (0) | 2 (2)
Psychiatric disorders NEC (Psychiatric disorders) | 2 (2) | 1 (1)
Renal disorder (Renal and urinary disorders) | 15 (16) | 7 (7)
Ureteric disorders (Renal and urinary disorders) | 3 (3) | 3 (3)
Pleural disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Skin and subcutaneous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bone and joint therapeutic procedures (Surgical and medical procedures) | 2 (3) | 0 (0)
Cardiac therapeutic procedures (Surgical and medical procedures) | 7 (7) | 10 (10)
Head and neck therapeutic procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal and urinary tract therapeutic procedures (Surgical and medical procedures) | 1 (2) | 0 (0)
Vascular therapeutic procedures (Surgical and medical procedures) | 1 (1) | 1 (1)
Aneurysms and artery dissections (Vascular disorders) | 4 (4) | 1 (1)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 6 (6) | 3 (3)
Vascular disorders NEC (Vascular disorders) | 4 (4) | 4 (4)
Vascular haemorrhagic disorders (Vascular disorders) | 4 (5) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=462) | Control Group (N=455)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Cardiac disorders) | 6 (6) | 8 (8)
Cardiac arrhythmias (Cardiac disorders) | 10 (12) | 10 (10)
Cardiac disorder signs and symptoms (Cardiac disorders) | 6 (6) | 4 (4)
Coronary artery disorders (Cardiac disorders) | 0 (0) | 2 (2)
Heart failures (Cardiac disorders) | 10 (17) | 19 (27)
Myocardial disorders (Cardiac disorders) | 0 (0) | 1 (1)
Hearing disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 1 (1)
Anterior eye structural change, deposit and degeneration (Eye disorders) | 2 (3) | 0 (0)
Infections - pathogen unspecified (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernias and other abdominal wall conditions (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 0 (0) | 2 (2)
Device issues (General disorders) | 1 (1) | 0 (0)
General system disorders NEC (General disorders) | 1 (1) | 6 (7)
Infections and infestations (Infections and infestations) | 0 (0) | 2 (2)
Bone and joint injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injuries NEC (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural and device related injuries and complications NEC (Injury, poisoning and procedural complications) | 17 (17) | 13 (15)
Cardiac and vascular investigations (excl enzyme tests) (Investigations) | 2 (2) | 3 (3)
Cardiac disorder signs and symptoms (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal investigations (Investigations) | 0 (0) | 1 (1)
Diabetic complications (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolism disorder (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorders (incl parkinsonism) (Nervous system disorders) | 0 (0) | 2 (2)
Neurological disorders NEC (Nervous system disorders) | 3 (3) | 8 (9)
Sleep disturbances (incl subtypes) (Nervous system disorders) | 1 (1) | 1 (1)
Renal disorder (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric disorders (Renal and urinary disorders) | 1 (1) | 4 (4)
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiac therapeutic procedures (Surgical and medical procedures) | 5 (5) | 7 (7)
Head and neck therapeutic procedures (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysms and artery dissections (Vascular disorders) | 1 (1) | 2 (2)
Decreased and nonspecific blood pressure disorders and shock (Surgical and medical procedures) | 0 (0) | 2 (2)
Vascular disorders NEC (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No